CLINICAL TRIAL: NCT00434512
Title: A Dose-ranging Study to Compare the Safety and Immunogenicity of a Candidate Human Deficiency Virus (HIV) Vaccine 732461, Adjuvanted or Not, Administered According to a 0, 1 Month Schedule to Healthy Adult HIV Seronegative Volunteers.
Brief Title: Dose-ranging Study to Evaluate the Safety & Immunogenicity of a HIV Vaccine 732461 in Healthy HIV Seronegative Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 108706; 2006-003796-12 (EudraCT Number)
Record Dates: First submitted 2007-02-12; First posted 2007-02-13 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: AIDS; HIV Infections
Keywords: Gag; vaccine; adjuvant; HIV; Pol; Nef
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- SB732461 adjuvanted_LD Group (Experimental): Healthy adult HIV seronegative subjects aged 18 to 40 years, who received two doses of the adjuvanted low-antigen dose [LD] (10 μg) SB732461 vaccine, intramuscularly, at Day 0 and Day 30.
  Interventions: Biological: HIV vaccine 732461
- SB732461 adjuvanted_MD Group (Experimental): Healthy adult HIV seronegative subjects aged 18 to 40 years, who received two doses of the adjuvanted medium-antigen dose [MD] (30 μg) SB732461 vaccine, intramuscularly, at Day 0 and Day 30.
  Interventions: Biological: HIV vaccine 732461
- SB732461 adjuvanted_HD Group (Experimental): Healthy adult HIV seronegative subjects aged 18 to 40 years, who received two doses of the adjuvanted high-antigen dose [HD] (90 μg) SB732461 vaccine, intramuscularly, at Day 0 and Day 30.
  Interventions: Biological: HIV vaccine 732461
- SB732461 non-adjuvanted_LD Group (Experimental): Healthy adult HIV seronegative subjects aged 18 to 40 years, who received two doses of the non-adjuvanted low-antigen dose [LD] (10 μg) SB732461 vaccine, intramuscularly, at Day 0 and Day 30.
  Interventions: Biological: HIV vaccine 732461
- SB732461 non-adjuvanted_MD Group (Experimental): Healthy adult HIV seronegative subjects aged 18 to 40 years, who received two doses of the non-adjuvanted medium-antigen dose [MD] (30 μg) SB732461 vaccine, intramuscularly, at Day 0 and Day 30.
  Interventions: Biological: HIV vaccine 732461
- SB732461 non-adjuvanted_HD Group (Experimental): Healthy adult HIV seronegative subjects aged 18 to 40 years, who received two doses of the non-adjuvanted high-antigen dose [HD] (90 μg) SB732461 vaccine, intramuscularly, at Day 0 and Day 30.
  Interventions: Biological: HIV vaccine 732461

INTERVENTIONS:
Biological: HIV vaccine 732461

SUMMARY:
GSK has constructed a new HIV immunogen comprised of conserved parts of the HIV virus (gag, pol and nef). The principal objectives of this study are to evaluate the reactogenicity and safety of this candidate vaccine with or without a GSK proprietary adjuvant system at three different doses and to evaluate the CD4+ T-cell response in terms of proportion of responders to the antigens two weeks after the second vaccination.

DETAILED DESCRIPTION:
This is a single center, observer-blind, randomized, dose-escalating, staggered study with 6 groups: 3 groups of 50 subjects receiving the adjuvanted candidate vaccine, at 3 different doses and 3 groups of 10 subjects receiving the non-adjuvanted candidate vaccine in water for injection, at 3 different doses. The vaccination schedule will be 0-1 month. Blood samples will be collected at 8 visits. The duration of the study will be approximately 14 months for each subject. Rationale for Protocol Posting Amendment: The third vaccination will be cancelled and the visit at Month 7 will be postponed to Month 9. The Protocol Posting has also been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* A male or female between and including 18-40 years at the time of first vaccination.
* Written informed consent obtained from the subject prior to any study procedure.
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* Good general health without significant medical history, physical examination findings, or clinically significant abnormal laboratory results.
* If the subject is female, she must be of non-childbearing potential, or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for 2 months after completion of the vaccination series.
* Negative for antibodies against HIV-1, HIV-2 and negative for HIV p24 antigen within 56 days (8 weeks) prior to enrolment. Subjects must be willing to accept HIV test results. Individuals who elect not to receive test results will not be enrolled.
* Negative for anti-HBc Ab, HBsAg and anti-HCV Ab.

Exclusion Criteria:

* Women who are pregnant or breast-feeding.
* Subjects with a history of, or current, alcohol or substance abuse.
* The subject is at high risk of acquiring HIV according to the behavioural risk assessment questionnaire.
* Morbid obesity
* Previous inclusion in a HIV vaccines trial.
* Receipt of live attenuated vaccines within 30 days of enrolment.
* Receipt of medically indicated subunit or killed vaccines or allergy treatment with antigen injections within 14 days of study vaccine administration.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Prior receipt of HIV-1 vaccines or placebo in a previous HIV vaccine trial.
* Receipt of blood products 120 days prior to HIV screening.
* Receipt of immunoglobulin 120 days prior to HIV screening.
* History of serious adverse reactions including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema and abdominal pain to vaccines.
* History of serious allergic reaction to any substance requiring hospitalization or emergency medical care.
* History of immunodeficiency or autoimmune disease.
* History of malignancy (unless there has been surgical excision followed by a sufficient observation period, of at least 5 years, to give a reasonable assurance of sustained cure and which, in the estimate of the investigator, is not likely to recur during the study period).
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccination.
* History of type I or type II diabetes mellitus including cases controlled with diet alone. A subject with past gestational diabetes is eligible.
* Thyroid disease including history of thyroidectomy and diagnoses requiring medication. A subject not requiring thyroid medicine within the past 12 months is eligible.
* Acute disease at the time of enrolment.
* Asthma requiring daily steroid or long acting β agonist prevention.
* Unstable asthma.
* Food- or wine-induced asthma.
* Known sensitivity to sulfites or aspirin.
* Bleeding disorder that was diagnosed by a physician. A subject who states that he or she has easy bruising or bleeding, but does not carry a formal diagnosis and has intramuscular (IM) injections and blood draws without any adverse experience is eligible.
* History of any serious neurologic disorder or seizure
* History of major congenital defect
* History of chronic fatigue syndrome or fibromyalgia
* Splenectomy
* Hypertension. A subject with hypertension is eligible if he or she is controlled on medication and the documented blood pressure is less than 150/100.
* Any medical, psychiatric or social condition, or occupational or other responsibility that, in the judgement of the investigator, would interfere with or serve as a contradiction to adherence to the study protocol or ability to give informed consent.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2007-02-20 (Actual); Primary Completion 2008-06-13 (Actual); Study Completion 2008-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below).
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Leroux-Roels G, Bourguignon P, Willekens J, Janssens M, Clement F, Didierlaurent AM, Fissette L, Roman F, Boutriau D. Immunogenicity and safety of a booster dose of an investigational adjuvanted polyprotein HIV-1 vaccine in healthy adults and effect of administration of chloroquine. Clin Vaccine Immunol. 2014 Mar;21(3):302-11. doi: 10.1128/CVI.00617-13. Epub 2014 Jan 3. PMID 24391139
- [Derived] Van Braeckel E, Koutsoukos M, Bourguignon P, Clement F, McNally L, Leroux-Roels G. Vaccine-induced HIV seropositivity: a problem on the rise. J Clin Virol. 2011 Apr;50(4):334-7. doi: 10.1016/j.jcv.2011.01.003. PMID 21300566
- [Derived] Van Braeckel E, Bourguignon P, Koutsoukos M, Clement F, Janssens M, Carletti I, Collard A, Demoitie MA, Voss G, Leroux-Roels G, McNally L. An adjuvanted polyprotein HIV-1 vaccine induces polyfunctional cross-reactive CD4+ T cell responses in seronegative volunteers. Clin Infect Dis. 2011 Feb 15;52(4):522-31. doi: 10.1093/cid/ciq160. Epub 2011 Jan 5. PMID 21208909

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 229 subjects were enrolled and screened in this study, and 49 of these were excluded before vaccination.
Period: Overall Study
Arm/Group | SB732461 Non-adjuvanted_LD Group | SB732461 Non-adjuvanted_MD Group | SB732461 Non-adjuvanted_HD Group | SB732461 adjuvanted_LD Group | SB732461 adjuvanted_MD Group | SB732461 adjuvanted_HD Group
Started | 10 | 10 | 10 | 50 | 50 | 50
Completed | 10 | 9 | 10 | 49 | 49 | 49
Not Completed | 0 | 1 | 0 | 1 | 1 | 1
Not completed — Migrated/moved from study area | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SB732461 Non-adjuvanted_LD Group | SB732461 Non-adjuvanted_MD Group | SB732461 Non-adjuvanted_HD Group | SB732461 adjuvanted_LD Group | SB732461 adjuvanted_MD Group | SB732461 adjuvanted_HD Group | Total
Number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 50 | 180
Age, Continuous [Mean (Standard Deviation); unit: Years] | 21.4 (3.75) | 21.8 (3.19) | 22.5 (4.99) | 22.0 (5.04) | 22.2 (3.66) | 22.9 (5.43) | 22.3 (4.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 7 | 33 | 28 | 32 | 114
  Male | 3 | 3 | 3 | 17 | 22 | 18 | 66
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Arabic/North African heritage | 1 | 0 | 0 | 0 | 1 | 0 | 2
  White - Caucasian/European heritage | 7 | 10 | 10 | 50 | 47 | 50 | 174
  Other - Unspecified | 2 | 0 | 0 | 0 | 2 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) follow-up period after each vaccination and overall (across doses)
Population: The analysis was performed on the Total Vaccinated Cohort, which included vaccinated subjects with at least one vaccine administration documented for whom data were available and who had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | SB732461 Non-adjuvanted_LD Group | SB732461 Non-adjuvanted_MD Group | SB732461 Non-adjuvanted_HD Group | SB732461 adjuvanted_LD Group | SB732461 adjuvanted_MD Group | SB732461 adjuvanted_HD Group
Number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 50
Participants
  Any Pain, Dose 1 | 2 | 0 | 2 | 49 | 49 | 49
  Grade 3 Pain, Dose 1 | 0 | 0 | 0 | 4 | 1 | 4
  Any Redness, Dose 1 | 0 | 0 | 0 | 5 | 18 | 9
  Grade 3 Redness, Dose 1 | 0 | 0 | 0 | 3 | 9 | 2
  Any Swelling, Dose 1 | 0 | 0 | 0 | 9 | 12 | 5
  Grade 3 Swelling, Dose 1 | 0 | 0 | 0 | 5 | 2 | 1
  Any Pain, Dose 2: number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 49
  Any Pain, Dose 2 | 3 | 2 | 4 | 47 | 49 | 48
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 49
  Grade 3 Pain, Dose 2 | 0 | 0 | 0 | 6 | 4 | 6
  Any Redness, Dose 2: number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 49
  Any Redness, Dose 2 | 0 | 0 | 0 | 14 | 17 | 25
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 49
  Grade 3 Redness, Dose 2 | 0 | 0 | 0 | 5 | 11 | 10
  Any Swelling, Dose 2: number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 49
  Any Swelling, Dose 2 | 0 | 0 | 0 | 11 | 13 | 17
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 49
  Grade 3 Swelling, Dose 2 | 0 | 0 | 0 | 4 | 2 | 3
  Any Pain, Overall | 3 | 2 | 5 | 49 | 50 | 50
  Grade 3 Pain, Overall | 0 | 0 | 0 | 7 | 5 | 10
  Any Redness, Overall | 0 | 0 | 0 | 14 | 23 | 25
  Grade 3 Redness, Overall | 0 | 0 | 0 | 7 | 13 | 12
  Any Swelling, Overall | 0 | 0 | 0 | 13 | 18 | 19
  Grade 3 Swelling, Overall | 0 | 0 | 0 | 6 | 3 | 4

2. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)], headache, myalgia, sweating, gastrointestinal symptoms(nausea, vomiting, diarrhea, and/or abdominal pain). Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) follow-up period after each vaccination and overall (across doses)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SB732461 Non-adjuvanted_LD Group | SB732461 Non-adjuvanted_MD Group | SB732461 Non-adjuvanted_HD Group | SB732461 adjuvanted_LD Group | SB732461 adjuvanted_MD Group | SB732461 adjuvanted_HD Group
Number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 50
Participants
  Any Fatigue, Dose 1 | 3 | 5 | 5 | 27 | 28 | 33
  Grade 3 Fatigue, Dose 1 | 0 | 0 | 0 | 2 | 0 | 1
  Related Fatigue, Dose 1 | 2 | 4 | 3 | 26 | 24 | 32
  Any Fever, Dose 1 | 0 | 0 | 0 | 3 | 3 | 3
  Grade 3 Fever, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  Related Fever, Dose 1 | 0 | 0 | 0 | 3 | 3 | 3
  Any Gastrointestinal, Dose 1 | 1 | 1 | 1 | 9 | 9 | 8
  Grade 3 Gastrointestinal, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  Related Gastrointestinal, Dose 1 | 1 | 0 | 1 | 8 | 6 | 5
  Any Headache, Dose 1 | 2 | 4 | 3 | 24 | 21 | 24
  Grade 3 Headache, Dose 1 | 0 | 0 | 0 | 2 | 0 | 2
  Related Headache, Dose 1 | 0 | 3 | 2 | 20 | 19 | 21
  Any Myalgia, Dose 1 | 2 | 1 | 1 | 13 | 20 | 23
  Grade 3 Myalgia, Dose 1 | 0 | 0 | 0 | 0 | 0 | 4
  Related Myalgia, Dose 1 | 2 | 1 | 1 | 13 | 19 | 21
  Any Sweating, Dose 1 | 0 | 0 | 2 | 7 | 8 | 11
  Grade 3 Sweating, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  Related Sweating, Dose 1 | 0 | 0 | 2 | 6 | 6 | 10
  Any Fatigue, Dose 2: number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 49
  Any Fatigue, Dose 2 | 3 | 2 | 4 | 39 | 43 | 44
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 49
  Grade 3 Fatigue, Dose 2 | 0 | 0 | 0 | 9 | 7 | 11
  Related Fatigue, Dose 2: number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 49
  Related Fatigue, Dose 2 | 3 | 1 | 3 | 39 | 43 | 44
  Any Fever, Dose 2: number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 49
  Any Fever, Dose 2 | 0 | 0 | 0 | 29 | 29 | 25
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 49
  Grade 3 Fever, Dose 2 | 0 | 0 | 0 | 3 | 2 | 1
  Related Fever, Dose 2: number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 49
  Related Fever, Dose 2 | 0 | 0 | 0 | 29 | 29 | 25
  Any Gastrointestinal, Dose 2: number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 49
  Any Gastrointestinal, Dose 2 | 1 | 1 | 2 | 20 | 15 | 13
  Grade 3 Gastrointestinal, Dose 2: number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 49
  Grade 3 Gastrointestinal, Dose 2 | 0 | 0 | 0 | 2 | 2 | 2
  Related Gastrointestinal, Dose 2: number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 49
  Related Gastrointestinal, Dose 2 | 1 | 1 | 2 | 19 | 12 | 11
  Any Headache, Dose 2: number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 49
  Any Headache, Dose 2 | 2 | 1 | 2 | 38 | 37 | 37
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 49
  Grade 3 Headache, Dose 2 | 0 | 0 | 0 | 8 | 5 | 6
  Related Headache, Dose 2: number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 49
  Related Headache, Dose 2 | 1 | 1 | 2 | 37 | 37 | 37
  Any Myalgia, Dose 2: number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 49
  Any Myalgia, Dose 2 | 0 | 1 | 1 | 31 | 31 | 28
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 49
  Grade 3 Myalgia, Dose 2 | 0 | 0 | 0 | 5 | 6 | 7
  Related Myalgia, Dose 2: number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 49
  Related Myalgia, Dose 2 | 0 | 1 | 1 | 31 | 31 | 28
  Any Sweating, Dose 2: number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 49
  Any Sweating, Dose 2 | 1 | 1 | 1 | 28 | 24 | 23
  Grade 3 Sweating, Dose 2: number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 49
  Grade 3 Sweating, Dose 2 | 0 | 0 | 0 | 3 | 2 | 4
  Related Sweating, Dose 2: number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 49
  Related Sweating, Dose 2 | 1 | 1 | 1 | 26 | 24 | 23
  Any Fatigue, Overall | 5 | 5 | 6 | 40 | 47 | 46
  Grade 3 Fatigue, Overall | 0 | 0 | 0 | 11 | 7 | 12
  Related Fatigue, Overall | 5 | 4 | 5 | 40 | 46 | 46
  Any Fever, Overall | 0 | 0 | 0 | 30 | 29 | 26
  Grade 3 Fever, Overall | 0 | 0 | 0 | 3 | 2 | 1
  Related Fever, Overall | 0 | 0 | 0 | 30 | 29 | 26
  Any Gastrointestinal, Overall | 2 | 2 | 2 | 23 | 21 | 17
  Grade 3 Gastrointestinal, Overall | 0 | 0 | 0 | 2 | 2 | 2
  Related Gastrointestinal, Overall | 2 | 1 | 2 | 22 | 16 | 13
  Any Headache, Overall | 4 | 4 | 5 | 42 | 42 | 41
  Grade 3 Headache, Overall | 0 | 0 | 0 | 10 | 5 | 8
  Related Headache, Overall | 1 | 3 | 4 | 40 | 42 | 41
  Any Myalgia, Overall | 2 | 1 | 2 | 31 | 35 | 36
  Grade 3 Myalgia, Overall | 0 | 0 | 0 | 5 | 6 | 8
  Related Myalgia, Overall | 2 | 1 | 2 | 31 | 35 | 35
  Any Sweating, Overall | 1 | 1 | 3 | 28 | 27 | 26
  Grade 3 Sweating, Overall | 0 | 0 | 0 | 3 | 2 | 4
  Related Sweating, Overall | 1 | 1 | 3 | 27 | 27 | 26

3. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 30-day (Days 0-29) follow-up period after vaccination (across doses)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SB732461 Non-adjuvanted_LD Group | SB732461 Non-adjuvanted_MD Group | SB732461 Non-adjuvanted_HD Group | SB732461 adjuvanted_LD Group | SB732461 adjuvanted_MD Group | SB732461 adjuvanted_HD Group
Number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 50
Participants
  Any AE(s) | 5 | 6 | 7 | 42 | 30 | 33
  Grade 3 AE(s) | 0 | 1 | 0 | 9 | 5 | 6
  Related AE(s) | 0 | 0 | 1 | 22 | 15 | 15

4. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs) and Related SAEs
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the whole study period (From Month 0 up to Month 12)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SB732461 Non-adjuvanted_LD Group | SB732461 Non-adjuvanted_MD Group | SB732461 Non-adjuvanted_HD Group | SB732461 adjuvanted_LD Group | SB732461 adjuvanted_MD Group | SB732461 adjuvanted_HD Group
Number analyzed (Participants) | 10 | 10 | 10 | 50 | 50 | 50
Participants
  SAEs: SAEs | 0 | 0 | 0 | 2 | 2 | 2
  Related SAEs: SAEs | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Subjects With Abnormal Haematological and Biochemical Levels at Month 0
Description: The frequency distribution of values below, within and above normal ranges, were tabulated per treatment group at each scheduled time point for the following biochemical or haematological parameters: red blood cells [RBC] count, haemoglobin, haematocrit, white blood cell [WBC] count, neutrophils, lymphocytes, monocytes, eosinophils, basophils, platelets, sodium, potassium, urea nitrogen, creatinine, alanine aminotransferase [ALT] and aspartate aminotransferase [AST].
Time Frame: At Month 0
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SB732461 Non-adjuvanted_LD Group | SB732461 adjuvanted_LD Group | SB732461 Non-adjuvanted_MD Group | SB732461 adjuvanted_MD Group | SB732461 Non-adjuvanted_HD Group | SB732461 adjuvanted_HD Group
Number analyzed (Participants) | 10 | 50 | 10 | 50 | 10 | 50
Participants
  RBC: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  RBC: Below | 0 | 2 | 1 | 1 | 1 | 2
  RBC: Within | 10 | 48 | 9 | 49 | 9 | 48
  RBC: Above | 0 | 0 | 0 | 0 | 0 | 0
  Haemoglobin: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Haemoglobin: Below | 0 | 4 | 1 | 0 | 0 | 1
  Haemoglobin: Within | 10 | 46 | 9 | 49 | 10 | 49
  Haemoglobin: Above | 0 | 0 | 0 | 1 | 0 | 0
  Hematocrit: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Hematocrit: Below | 0 | 3 | 1 | 1 | 1 | 2
  Hematocrit: Within | 10 | 47 | 9 | 49 | 9 | 48
  Hematocrit: Above | 0 | 0 | 0 | 0 | 0 | 0
  WBC: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  WBC: Below | 1 | 1 | 0 | 4 | 0 | 6
  WBC: Within | 9 | 47 | 10 | 45 | 10 | 44
  WBC: Above | 0 | 2 | 0 | 1 | 0 | 0
  Neutrophils: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils: Below | 0 | 2 | 0 | 2 | 0 | 3
  Neutrophils: Within | 9 | 43 | 10 | 46 | 10 | 47
  Neutrophils: Above | 1 | 5 | 0 | 2 | 0 | 0
  Lymphocytes: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Below | 1 | 6 | 0 | 2 | 0 | 0
  Lymphocytes: Within | 9 | 44 | 10 | 46 | 10 | 48
  Lymphocytes: Above | 0 | 0 | 0 | 2 | 0 | 2
  Monocytes: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes: Below | 0 | 3 | 0 | 0 | 0 | 0
  Monocytes: Within | 9 | 40 | 7 | 40 | 7 | 39
  Monocytes: Above | 1 | 7 | 3 | 10 | 3 | 11
  Eosinophils: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils: Below | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils: Within | 7 | 47 | 9 | 49 | 10 | 49
  Eosinophils: Above | 3 | 3 | 1 | 1 | 0 | 1
  Basophils: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Basophils: Below | 0 | 0 | 0 | 0 | 0 | 0
  Basophils: Within | 10 | 50 | 10 | 50 | 10 | 50
  Basophils: Above | 0 | 0 | 0 | 0 | 0 | 0
  Platelets: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Platelets: Below | 1 | 0 | 0 | 2 | 1 | 1
  Platelets: Within | 9 | 50 | 10 | 48 | 9 | 49
  Platelets: Above | 0 | 0 | 0 | 0 | 0 | 0
  Sodium: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Sodium: Below | 0 | 0 | 0 | 0 | 0 | 0
  Sodium: Within | 10 | 49 | 10 | 50 | 10 | 50
  Sodium: Above | 0 | 1 | 0 | 0 | 0 | 0
  Potassium: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Potassium: Below | 0 | 2 | 0 | 0 | 0 | 0
  Potassium: Within | 10 | 48 | 10 | 49 | 9 | 50
  Potassium: Above | 0 | 0 | 0 | 1 | 1 | 0
  Urea Nitrogen: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Urea Nitrogen: Below | 0 | 0 | 0 | 0 | 0 | 0
  Urea Nitrogen: Within | 10 | 49 | 10 | 50 | 10 | 50
  Urea Nitrogen: Above | 0 | 1 | 0 | 0 | 0 | 0
  Creatinine: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine: Below | 0 | 0 | 0 | 1 | 0 | 0
  Creatinine: Within | 10 | 49 | 9 | 48 | 10 | 49
  Creatinine: Above | 0 | 1 | 1 | 1 | 0 | 1
  AST: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  AST: Below | 0 | 0 | 0 | 0 | 0 | 0
  AST: Within | 10 | 50 | 10 | 48 | 10 | 49
  AST: Above | 0 | 0 | 0 | 2 | 0 | 1
  ALT: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  ALT: Below | 0 | 2 | 0 | 0 | 0 | 0
  ALT: Within | 10 | 48 | 10 | 50 | 10 | 49
  ALT: Above | 0 | 0 | 0 | 0 | 0 | 1

6. Primary Outcome: Number of Subjects With Abnormal Haematological and Biochemical Levels at Month 1
Description: as for outcome 5
Time Frame: At Month 1
Population: The analysis was preformed on the Total Vaccinated cohort, which included vaccinated subjects with at least one vaccine administration documented for whom data were available and who had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | SB732461 Non-adjuvanted_LD Group | SB732461 adjuvanted_LD Group | SB732461 Non-adjuvanted_MD Group | SB732461 adjuvanted_MD Group | SB732461 Non-adjuvanted_HD Group | SB732461 adjuvanted_HD Group
Number analyzed (Participants) | 10 | 50 | 10 | 50 | 10 | 50
Participants
  RBC: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  RBC: Below | 0 | 0 | 0 | 0 | 0 | 0
  RBC: Within | 10 | 50 | 10 | 50 | 10 | 49
  RBC: Above | 0 | 0 | 0 | 0 | 0 | 1
  Haemoglobin: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Haemoglobin: Below | 0 | 2 | 0 | 1 | 0 | 0
  Haemoglobin: Within | 10 | 48 | 10 | 49 | 10 | 50
  Haemoglobin: Above | 0 | 0 | 0 | 0 | 0 | 0
  Hematocrit: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Hematocrit: Below | 0 | 4 | 0 | 1 | 0 | 0
  Hematocrit: Within | 10 | 46 | 10 | 49 | 10 | 50
  Hematocrit: Above | 0 | 0 | 0 | 0 | 0 | 0
  WBC: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  WBC: Below | 0 | 1 | 0 | 7 | 0 | 4
  WBC: Within | 10 | 48 | 10 | 42 | 10 | 45
  WBC: Above | 0 | 1 | 0 | 1 | 0 | 1
  Neutrophils: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils: Below | 0 | 2 | 1 | 5 | 0 | 4
  Neutrophils: Within | 10 | 46 | 9 | 44 | 10 | 43
  Neutrophils: Above | 0 | 2 | 0 | 1 | 0 | 3
  Lymphocytes: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Below | 0 | 2 | 0 | 0 | 0 | 3
  Lymphocytes: Within | 10 | 47 | 9 | 47 | 10 | 43
  Lymphocytes: Above | 0 | 1 | 1 | 3 | 0 | 4
  Monocytes: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes: Below | 0 | 1 | 0 | 0 | 0 | 0
  Monocytes: Within | 7 | 38 | 6 | 39 | 5 | 31
  Monocytes: Above | 3 | 11 | 4 | 11 | 5 | 19
  Eosinophils: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils: Below | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils: Within | 9 | 44 | 9 | 44 | 10 | 47
  Eosinophils: Above | 1 | 6 | 1 | 6 | 0 | 3
  Basophils: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Basophils: Below | 0 | 0 | 0 | 0 | 0 | 0
  Basophils: Within | 10 | 50 | 10 | 50 | 10 | 50
  Basophils: Above | 0 | 0 | 0 | 0 | 0 | 0
  Platelets: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Platelets: Below | 0 | 0 | 0 | 0 | 1 | 2
  Platelets: Within | 10 | 50 | 10 | 50 | 9 | 48
  Platelets: Above | 0 | 0 | 0 | 0 | 0 | 0
  Sodium: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Sodium: Below | 0 | 0 | 0 | 0 | 0 | 0
  Sodium: Within | 10 | 50 | 10 | 48 | 9 | 49
  Sodium: Above | 0 | 0 | 0 | 2 | 1 | 1
  Potassium: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Potassium: Below | 0 | 1 | 0 | 0 | 0 | 0
  Potassium: Within | 10 | 47 | 10 | 47 | 10 | 45
  Potassium: Above | 0 | 2 | 0 | 3 | 0 | 5
  Urea Nitrogen: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Urea Nitrogen: Below | 0 | 0 | 0 | 0 | 0 | 0
  Urea Nitrogen: Within | 10 | 49 | 9 | 50 | 10 | 49
  Urea Nitrogen: Above | 0 | 1 | 1 | 0 | 0 | 1
  Creatinine: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine: Below | 0 | 0 | 0 | 1 | 0 | 0
  Creatinine: Within | 10 | 48 | 10 | 48 | 10 | 50
  Creatinine: Above | 0 | 2 | 0 | 1 | 0 | 0
  AST: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  AST: Below | 0 | 0 | 0 | 0 | 0 | 0
  AST: Within | 10 | 49 | 10 | 49 | 10 | 47
  AST: Above | 0 | 1 | 0 | 1 | 0 | 3
  ALT: Unknown | 0 | 0 | 0 | 0 | 0 | 0
  ALT: Below | 0 | 1 | 0 | 1 | 0 | 0
  ALT: Within | 10 | 49 | 10 | 48 | 10 | 47
  ALT: Above | 0 | 0 | 0 | 1 | 0 | 3

7. Primary Outcome: Number of Subjects With Abnormal Haematological and Biochemical Levels at Day 44
Description: as for outcome 5
Time Frame: At Day 44
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | SB732461 Non-adjuvanted_LD Group | SB732461 adjuvanted_LD Group | SB732461 Non-adjuvanted_MD Group | SB732461 adjuvanted_MD Group | SB732461 Non-adjuvanted_HD Group | SB732461 adjuvanted_HD Group
Number analyzed (Participants) | 10 | 50 | 10 | 50 | 10 | 50
Participants
  RBC: Unknown | 0 | 0 | 0 | 0 | 0 | 2
  RBC: Below | 0 | 0 | 0 | 1 | 0 | 1
  RBC: Within | 10 | 50 | 10 | 49 | 10 | 47
  RBC: Above | 0 | 0 | 0 | 0 | 0 | 0
  Haemoglobin: Unknown | 0 | 0 | 0 | 0 | 0 | 2
  Haemoglobin: Below | 1 | 1 | 0 | 2 | 2 | 2
  Haemoglobin: Within | 9 | 49 | 10 | 48 | 8 | 46
  Haemoglobin: Above | 0 | 0 | 0 | 0 | 0 | 0
  Hematocrit: Unknown | 0 | 0 | 0 | 0 | 0 | 2
  Hematocrit: Below | 1 | 2 | 0 | 2 | 2 | 4
  Hematocrit: Within | 9 | 48 | 10 | 48 | 8 | 44
  Hematocrit: Above | 0 | 0 | 0 | 0 | 0 | 0
  WBC: Unknown | 0 | 0 | 0 | 0 | 0 | 2
  WBC: Below | 1 | 0 | 1 | 4 | 0 | 0
  WBC: Within | 9 | 48 | 9 | 46 | 10 | 47
  WBC: Above | 0 | 2 | 0 | 0 | 0 | 1
  Neutrophils: Unknown | 0 | 0 | 0 | 0 | 0 | 2
  Neutrophils: Below | 0 | 2 | 1 | 3 | 1 | 1
  Neutrophils: Within | 10 | 47 | 9 | 47 | 8 | 46
  Neutrophils: Above | 0 | 1 | 0 | 0 | 1 | 1
  Lymphocytes: Unknown | 0 | 0 | 0 | 0 | 0 | 2
  Lymphocytes: Below | 0 | 2 | 0 | 0 | 1 | 2
  Lymphocytes: Within | 10 | 46 | 9 | 47 | 8 | 45
  Lymphocytes: Above | 0 | 2 | 1 | 3 | 1 | 1
  Monocytes: Unknown | 0 | 0 | 0 | 0 | 0 | 2
  Monocytes: Below | 1 | 0 | 0 | 0 | 0 | 2
  Monocytes: Within | 6 | 44 | 7 | 42 | 6 | 34
  Monocytes: Above | 3 | 6 | 3 | 8 | 4 | 12
  Eosinophils: Unknown | 0 | 0 | 0 | 0 | 0 | 2
  Eosinophils: Below | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils: Within | 8 | 46 | 9 | 46 | 10 | 47
  Eosinophils: Above | 2 | 4 | 1 | 4 | 0 | 1
  Basophils: Unknown | 0 | 0 | 0 | 0 | 0 | 2
  Basophils: Below | 0 | 0 | 0 | 0 | 0 | 0
  Basophils: Within | 10 | 50 | 10 | 50 | 10 | 48
  Basophils: Above | 0 | 0 | 0 | 0 | 0 | 0
  Platelets: Unknown | 0 | 0 | 0 | 0 | 0 | 2
  Platelets: Below | 0 | 0 | 0 | 0 | 0 | 1
  Platelets: Within | 10 | 50 | 10 | 50 | 10 | 47
  Platelets: Above | 0 | 0 | 0 | 0 | 0 | 0
  Sodium: Unknown | 0 | 0 | 0 | 0 | 0 | 2
  Sodium: Below | 0 | 0 | 0 | 0 | 0 | 0
  Sodium: Within | 9 | 50 | 10 | 50 | 10 | 48
  Sodium: Above | 1 | 0 | 0 | 0 | 0 | 0
  Potassium: Unknown | 0 | 0 | 0 | 0 | 0 | 2
  Potassium: Below | 0 | 0 | 0 | 0 | 0 | 1
  Potassium: Within | 10 | 48 | 10 | 49 | 10 | 46
  Potassium: Above | 0 | 2 | 0 | 1 | 0 | 1
  Urea Nitrogen: Unknown | 0 | 0 | 0 | 0 | 0 | 2
  Urea Nitrogen: Below | 0 | 0 | 0 | 0 | 0 | 0
  Urea Nitrogen: Within | 10 | 48 | 10 | 49 | 10 | 47
  Urea Nitrogen: Above | 0 | 2 | 0 | 1 | 0 | 1
  Creatinine: Unknown | 0 | 0 | 0 | 0 | 0 | 2
  Creatinine: Below | 1 | 0 | 0 | 0 | 1 | 2
  Creatinine: Within | 9 | 47 | 10 | 50 | 9 | 43
  Creatinine: Above | 0 | 3 | 0 | 0 | 0 | 3
  AST: Unknown | 0 | 0 | 0 | 0 | 0 | 2
  AST: Below | 0 | 0 | 0 | 0 | 0 | 0
  AST: Within | 10 | 50 | 10 | 49 | 10 | 48
  AST: Above | 0 | 0 | 0 | 1 | 0 | 0
  ALT: Unknown | 0 | 0 | 0 | 0 | 0 | 2
  ALT: Below | 0 | 1 | 0 | 0 | 0 | 1
  ALT: Within | 10 | 48 | 10 | 49 | 10 | 47
  ALT: Above | 0 | 1 | 0 | 1 | 0 | 0

8. Primary Outcome: Number of Subjects With Abnormal Haematological and Biochemical Levels at Month 2
Description: The frequency distribution of values below, within and above normal ranges, were tabulated per treatment group at each scheduled time point for the following biochemical or haematological parameters: red blood cells [RBC] count, haemoglobin, haematocrit, white blood cell [RBC] count, neutrophils, lymphocytes, monocytes, eosinophils, basophils, platelets, sodium, potassium, urea nitrogen, creatinine, alanine aminotransferase [ALT] and aspartate aminotransferase [AST].
Time Frame: At Month 2
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | SB732461 Non-adjuvanted_LD Group | SB732461 adjuvanted_LD Group | SB732461 Non-adjuvanted_MD Group | SB732461 adjuvanted_MD Group | SB732461 Non-adjuvanted_HD Group | SB732461 adjuvanted_HD Group
Number analyzed (Participants) | 10 | 50 | 10 | 50 | 10 | 50
Participants
  RBC: Unknown | 0 | 0 | 0 | 1 | 0 | 1
  RBC: Below | 0 | 0 | 1 | 1 | 0 | 0
  RBC: Within | 10 | 50 | 9 | 48 | 10 | 49
  RBC: Above | 0 | 0 | 0 | 0 | 0 | 0
  Haemoglobin: Unknown | 0 | 0 | 0 | 1 | 0 | 1
  Haemoglobin: Below | 1 | 3 | 1 | 2 | 1 | 1
  Haemoglobin: Within | 9 | 47 | 9 | 47 | 9 | 48
  Haemoglobin: Above | 0 | 0 | 0 | 0 | 0 | 0
  Hematocrit: Unknown | 0 | 0 | 0 | 1 | 0 | 1
  Hematocrit: Below | 1 | 3 | 1 | 1 | 1 | 0
  Hematocrit: Within | 9 | 47 | 9 | 48 | 9 | 49
  Hematocrit: Above | 0 | 0 | 0 | 0 | 0 | 0
  WBC: Unknown | 0 | 0 | 0 | 1 | 0 | 1
  WBC: Below | 2 | 1 | 0 | 5 | 1 | 5
  WBC: Within | 8 | 48 | 10 | 43 | 9 | 43
  WBC: Above | 0 | 1 | 0 | 1 | 0 | 1
  Neutrophils: Unknown | 0 | 0 | 0 | 1 | 0 | 1
  Neutrophils: Below | 1 | 3 | 1 | 4 | 0 | 5
  Neutrophils: Within | 9 | 45 | 9 | 45 | 10 | 42
  Neutrophils: Above | 0 | 2 | 0 | 0 | 0 | 2
  Lymphocytes: Unknown | 0 | 0 | 0 | 1 | 0 | 1
  Lymphocytes: Below | 0 | 2 | 0 | 1 | 0 | 3
  Lymphocytes: Within | 10 | 48 | 9 | 43 | 10 | 42
  Lymphocytes: Above | 0 | 0 | 1 | 5 | 0 | 4
  Monocytes: Unknown | 0 | 0 | 0 | 1 | 0 | 1
  Monocytes: Below | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes: Within | 6 | 43 | 5 | 37 | 9 | 33
  Monocytes: Above | 4 | 7 | 5 | 12 | 1 | 16
  Eosinophils: Unknown | 0 | 0 | 0 | 1 | 0 | 1
  Eosinophils: Below | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils: Within | 7 | 47 | 9 | 41 | 10 | 46
  Eosinophils: Above | 3 | 3 | 1 | 8 | 0 | 3
  Basophils: Unknown | 0 | 0 | 0 | 1 | 0 | 1
  Basophils: Below | 0 | 0 | 0 | 0 | 0 | 0
  Basophils: Within | 10 | 50 | 10 | 49 | 10 | 49
  Basophils: Above | 0 | 0 | 0 | 0 | 0 | 0
  Platelets: Unknown | 0 | 0 | 0 | 1 | 0 | 1
  Platelets: Below | 0 | 2 | 0 | 0 | 1 | 1
  Platelets: Within | 10 | 48 | 10 | 48 | 9 | 48
  Platelets: Above | 0 | 0 | 0 | 1 | 0 | 0
  Sodium: Unknown | 0 | 0 | 0 | 1 | 0 | 1
  Sodium: Below | 0 | 0 | 0 | 0 | 1 | 0
  Sodium: Within | 10 | 50 | 9 | 48 | 9 | 49
  Sodium: Above | 0 | 0 | 1 | 1 | 0 | 0
  Potassium: Unknown | 0 | 0 | 0 | 1 | 0 | 1
  Potassium: Below | 0 | 0 | 0 | 1 | 1 | 0
  Potassium: Within | 10 | 50 | 10 | 48 | 9 | 49
  Potassium: Above | 0 | 0 | 0 | 0 | 0 | 0
  Urea Nitrogen: Unknown | 0 | 0 | 0 | 1 | 0 | 1
  Urea Nitrogen: Below | 0 | 0 | 0 | 0 | 0 | 0
  Urea Nitrogen: Within | 9 | 48 | 10 | 48 | 10 | 48
  Urea Nitrogen: Above | 1 | 2 | 0 | 1 | 0 | 1
  Creatinine: Unknown | 0 | 0 | 0 | 1 | 0 | 1
  Creatinine: Below | 1 | 0 | 0 | 1 | 0 | 1
  Creatinine: Within | 9 | 49 | 10 | 48 | 10 | 47
  Creatinine: Above | 0 | 1 | 0 | 0 | 0 | 1
  AST: Unknown | 0 | 0 | 0 | 1 | 0 | 1
  AST: Below | 0 | 0 | 0 | 0 | 0 | 0
  AST: Within | 10 | 50 | 10 | 48 | 10 | 49
  AST: Above | 0 | 0 | 0 | 1 | 0 | 0
  ALT: Unknown | 0 | 0 | 0 | 1 | 0 | 1
  ALT: Below | 0 | 1 | 0 | 0 | 0 | 0
  ALT: Within | 10 | 48 | 10 | 48 | 10 | 48
  ALT: Above | 0 | 1 | 0 | 1 | 0 | 1

9. Primary Outcome: Number of Subjects With Abnormal Haematological and Biochemical Levels at Month 6
Description: as for outcome 5
Time Frame: At Month 6
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | SB732461 Non-adjuvanted_LD Group | SB732461 adjuvanted_LD Group | SB732461 Non-adjuvanted_MD Group | SB732461 adjuvanted_MD Group | SB732461 Non-adjuvanted_HD Group | SB732461 adjuvanted_HD Group
Number analyzed (Participants) | 10 | 50 | 10 | 50 | 10 | 50
Participants
  Haemoglobin: Unknwon | 0 | 1 | 1 | 1 | 2 | 2
  Haemoglobin: Below | 0 | 1 | 0 | 2 | 0 | 1
  Haemoglobin: Within | 10 | 48 | 9 | 47 | 8 | 47
  Haemoglobin: Above | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes: Unknwon | 0 | 1 | 1 | 1 | 2 | 2
  Monocytes: Below | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes: Within | 8 | 41 | 7 | 34 | 6 | 30
  Monocytes: Above | 2 | 8 | 2 | 15 | 2 | 18
  Sodium: Unknwon | 0 | 1 | 1 | 1 | 2 | 1
  Sodium: Below | 0 | 0 | 0 | 0 | 0 | 0
  Sodium: Within | 10 | 49 | 9 | 48 | 8 | 49
  Sodium: Above | 0 | 0 | 0 | 1 | 0 | 0
  Potassium: Unknwon | 0 | 1 | 1 | 1 | 2 | 1
  Potassium: Below | 0 | 0 | 0 | 0 | 1 | 1
  Potassium: Within | 10 | 49 | 9 | 49 | 7 | 47
  Potassium: Above | 0 | 0 | 0 | 0 | 0 | 1
  RBC: Unknwon | 0 | 1 | 1 | 1 | 2 | 2
  RBC: Below | 0 | 1 | 0 | 0 | 0 | 0
  RBC: Within | 10 | 48 | 9 | 49 | 8 | 47
  RBC: Above | 0 | 0 | 0 | 0 | 0 | 1
  Lymphocytes: Unknwon | 0 | 1 | 1 | 1 | 2 | 2
  Lymphocytes: Below | 0 | 1 | 1 | 0 | 0 | 0
  Lymphocytes: Within | 10 | 48 | 8 | 44 | 8 | 44
  Lymphocytes: Above | 0 | 0 | 0 | 5 | 0 | 4
  Platelets: Unknwon | 0 | 1 | 1 | 1 | 2 | 2
  Platelets: Below | 0 | 0 | 0 | 1 | 0 | 3
  Platelets: Within | 10 | 49 | 9 | 48 | 8 | 45
  Platelets: Above | 0 | 0 | 0 | 0 | 0 | 0
  Urea Nitrogen: Unknwon | 0 | 1 | 1 | 1 | 2 | 1
  Urea Nitrogen: Below | 0 | 0 | 0 | 0 | 0 | 0
  Urea Nitrogen: Within | 10 | 48 | 9 | 49 | 8 | 49
  Urea Nitrogen: Above | 0 | 1 | 0 | 0 | 0 | 0
  Hematocrit: Unknwon | 0 | 1 | 1 | 1 | 2 | 2
  Hematocrit: Below | 1 | 1 | 1 | 2 | 0 | 2
  Hematocrit: Within | 9 | 48 | 8 | 47 | 8 | 46
  Hematocrit: Above | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine: Unknwon | 0 | 1 | 1 | 1 | 2 | 1
  Creatinine: Below | 0 | 0 | 0 | 0 | 0 | 1
  Creatinine: Within | 10 | 49 | 8 | 48 | 8 | 46
  Creatinine: Above | 0 | 0 | 1 | 1 | 0 | 2
  AST: Unknwon | 0 | 1 | 1 | 1 | 2 | 1
  AST: Below | 0 | 0 | 0 | 0 | 0 | 0
  AST: Within | 10 | 48 | 9 | 49 | 8 | 49
  AST: Above | 0 | 1 | 0 | 0 | 0 | 0
  ALT: Unknwon | 0 | 1 | 1 | 1 | 2 | 1
  ALT: Below | 0 | 1 | 0 | 0 | 1 | 0
  ALT: Within | 10 | 46 | 9 | 49 | 7 | 48
  ALT: Above | 0 | 2 | 0 | 0 | 0 | 1
  Neutrophils: Unknwon | 0 | 1 | 1 | 1 | 2 | 2
  Neutrophils: Below | 0 | 1 | 0 | 6 | 0 | 4
  Neutrophils: Within | 10 | 48 | 8 | 43 | 8 | 44
  Neutrophils: Above | 0 | 0 | 1 | 0 | 0 | 0
  Basophils: Unknwon | 0 | 1 | 1 | 1 | 2 | 2
  Basophils: Below | 0 | 0 | 0 | 0 | 0 | 0
  Basophils: Within | 10 | 49 | 9 | 49 | 8 | 48
  Basophils: Above | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils: Unknwon | 0 | 1 | 1 | 1 | 2 | 2
  Eosinophils: Below | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils: Within | 9 | 46 | 8 | 42 | 8 | 48
  Eosinophils: Above | 1 | 3 | 1 | 7 | 0 | 0
  WBC: Unknwon | 0 | 1 | 1 | 1 | 2 | 2
  WBC: Below | 1 | 2 | 0 | 7 | 0 | 3
  WBC: Within | 9 | 47 | 9 | 42 | 8 | 42
  WBC: Above | 0 | 0 | 0 | 0 | 0 | 3

10. Primary Outcome: Number of Subjects With Abnormal Haematological and Biochemical Levels at Month 9
Description: as for outcome 5
Time Frame: At Month 9
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | SB732461 Non-adjuvanted_LD Group | SB732461 adjuvanted_LD Group | SB732461 Non-adjuvanted_MD Group | SB732461 adjuvanted_MD Group | SB732461 Non-adjuvanted_HD Group | SB732461 adjuvanted_HD Group
Number analyzed (Participants) | 10 | 50 | 10 | 50 | 10 | 50
Participants
  Haemoglobin: Unknown | 0 | 1 | 0 | 0 | 1 | 2
  Haemoglobin: Below | 0 | 1 | 0 | 0 | 0 | 3
  Haemoglobin: Within | 10 | 47 | 10 | 50 | 9 | 45
  Haemoglobin: Above | 0 | 1 | 0 | 0 | 0 | 0
  Monocytes: Unknown | 0 | 1 | 0 | 0 | 1 | 2
  Monocytes: Below | 0 | 0 | 0 | 1 | 0 | 0
  Monocytes: Within | 8 | 32 | 8 | 38 | 6 | 35
  Monocytes: Above | 2 | 17 | 2 | 11 | 3 | 13
  Sodium: Unknown | 0 | 1 | 0 | 0 | 1 | 2
  Sodium: Below | 0 | 0 | 0 | 0 | 0 | 0
  Sodium: Within | 10 | 49 | 10 | 50 | 9 | 46
  Sodium: Above | 0 | 0 | 0 | 0 | 0 | 2
  Potassium: Unknown | 0 | 1 | 0 | 0 | 1 | 2
  Potassium: Below | 0 | 0 | 0 | 0 | 0 | 0
  Potassium: Within | 9 | 46 | 10 | 48 | 9 | 48
  Potassium: Above | 1 | 3 | 0 | 2 | 0 | 0
  RBC: Unknown | 0 | 1 | 0 | 0 | 1 | 2
  RBC: Below | 0 | 0 | 0 | 0 | 0 | 1
  RBC: Within | 10 | 49 | 10 | 50 | 9 | 46
  RBC: Above | 0 | 0 | 0 | 0 | 0 | 1
  Lymphocytes: Unknown | 0 | 1 | 0 | 0 | 1 | 2
  Lymphocytes: Below | 0 | 1 | 1 | 3 | 0 | 3
  Lymphocytes: Within | 9 | 46 | 9 | 47 | 9 | 44
  Lymphocytes: Above | 1 | 2 | 0 | 0 | 0 | 1
  Platelets: Unknown | 0 | 1 | 0 | 0 | 1 | 2
  Platelets: Below | 1 | 0 | 0 | 0 | 0 | 0
  Platelets: Within | 9 | 48 | 10 | 50 | 9 | 48
  Platelets: Above | 0 | 1 | 0 | 0 | 0 | 0
  Urea Nitrogen: Unknown | 0 | 1 | 0 | 0 | 1 | 2
  Urea Nitrogen: Below | 0 | 0 | 0 | 0 | 0 | 0
  Urea Nitrogen: Within | 10 | 49 | 10 | 49 | 8 | 47
  Urea Nitrogen: Above | 0 | 0 | 0 | 1 | 1 | 1
  Hematocrit: Unknown | 0 | 1 | 0 | 0 | 1 | 2
  Hematocrit: Below | 0 | 3 | 0 | 0 | 0 | 3
  Hematocrit: Within | 10 | 46 | 10 | 50 | 9 | 45
  Hematocrit: Above | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine: Unknown | 0 | 1 | 0 | 0 | 1 | 2
  Creatinine: Below | 0 | 0 | 0 | 0 | 0 | 3
  Creatinine: Within | 10 | 48 | 10 | 50 | 9 | 45
  Creatinine: Above | 0 | 1 | 0 | 0 | 0 | 0
  AST: Unknown | 0 | 1 | 0 | 0 | 1 | 2
  AST: Below | 0 | 0 | 0 | 0 | 0 | 0
  AST: Within | 10 | 48 | 10 | 50 | 9 | 46
  AST: Above | 0 | 1 | 0 | 0 | 0 | 2
  ALT: Unknown | 0 | 1 | 0 | 0 | 1 | 2
  ALT: Below | 0 | 0 | 0 | 1 | 0 | 1
  ALT: Within | 10 | 48 | 10 | 49 | 9 | 45
  ALT: Above | 0 | 1 | 0 | 0 | 0 | 2
  Neutrophils: Unknown | 0 | 1 | 0 | 0 | 1 | 2
  Neutrophils: Below | 2 | 2 | 0 | 2 | 0 | 1
  Neutrophils: Within | 8 | 46 | 10 | 46 | 9 | 47
  Neutrophils: Above | 0 | 1 | 0 | 2 | 0 | 0
  Basophils: Unknown | 0 | 1 | 0 | 0 | 1 | 2
  Basophils: Below | 0 | 0 | 0 | 0 | 0 | 0
  Basophils: Within | 10 | 49 | 10 | 50 | 9 | 48
  Basophils: Above | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils: Unknown | 0 | 1 | 0 | 0 | 1 | 2
  Eosinophils: Below | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils: Within | 8 | 45 | 10 | 46 | 9 | 48
  Eosinophils: Above | 2 | 4 | 0 | 4 | 0 | 0
  WBC: Unknown | 0 | 1 | 0 | 0 | 1 | 2
  WBC: Below | 0 | 3 | 0 | 2 | 0 | 3
  WBC: Within | 10 | 46 | 9 | 47 | 9 | 43
  WBC: Above | 0 | 0 | 1 | 1 | 0 | 2

11. Primary Outcome: Number of Subjects With Abnormal Haematological and Biochemical Levels at Month 12
Description: as for outcome 5
Time Frame: At Month 12
Population: The analysis was preformed on the Total Vaccinated cohort, which included vaccinated subjects with at least one vaccination administration documented for whom data were available and who had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | SB732461 Non-adjuvanted_LD Group | SB732461 adjuvanted_LD Group | SB732461 Non-adjuvanted_MD Group | SB732461 adjuvanted_MD Group | SB732461 Non-adjuvanted_HD Group | SB732461 adjuvanted_HD Group
Number analyzed (Participants) | 10 | 50 | 10 | 50 | 10 | 50
Participants
  Haemoglobin: Unknown | 0 | 1 | 1 | 1 | 0 | 1
  Haemoglobin: Below | 0 | 2 | 1 | 2 | 0 | 0
  Haemoglobin: Whitin | 10 | 47 | 8 | 47 | 10 | 49
  Haemoglobin: Above | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes: Unknown | 0 | 1 | 1 | 1 | 0 | 1
  Monocytes: Below | 0 | 0 | 0 | 1 | 0 | 0
  Monocytes: Whitin | 8 | 45 | 6 | 38 | 8 | 41
  Monocytes: Above | 2 | 4 | 3 | 10 | 2 | 8
  Sodium: Unknown | 0 | 1 | 1 | 1 | 0 | 1
  Sodium: Below | 0 | 0 | 0 | 0 | 0 | 0
  Sodium: Whitin | 10 | 45 | 9 | 44 | 10 | 49
  Sodium: Above | 0 | 4 | 0 | 5 | 0 | 0
  Potassium: Unknown | 0 | 1 | 1 | 1 | 0 | 1
  Potassium: Below | 1 | 1 | 0 | 1 | 1 | 0
  Potassium: Whitin | 9 | 48 | 9 | 48 | 9 | 49
  Potassium: Above | 0 | 0 | 0 | 0 | 0 | 0
  RBC: Unknown | 0 | 1 | 1 | 1 | 0 | 1
  RBC: Below | 0 | 0 | 0 | 1 | 0 | 1
  RBC: Whitin | 10 | 49 | 9 | 48 | 10 | 47
  RBC: Above | 0 | 0 | 0 | 0 | 0 | 1
  Lymphocytes: Unknown | 0 | 1 | 1 | 1 | 0 | 1
  Lymphocytes: Below | 0 | 3 | 1 | 0 | 0 | 2
  Lymphocytes: Whitin | 10 | 43 | 7 | 43 | 10 | 45
  Lymphocytes: Above | 0 | 3 | 1 | 6 | 0 | 2
  Platelets: Unknown | 0 | 1 | 1 | 1 | 0 | 1
  Platelets: Below | 1 | 0 | 0 | 0 | 0 | 0
  Platelets: Whitin | 9 | 49 | 9 | 49 | 10 | 49
  Platelets: Above | 0 | 0 | 0 | 0 | 0 | 0
  Urea Nitrogen: Unknown | 0 | 1 | 1 | 1 | 0 | 1
  Urea Nitrogen: Below | 0 | 0 | 0 | 0 | 0 | 0
  Urea Nitrogen: Whitin | 10 | 46 | 7 | 49 | 10 | 48
  Urea Nitrogen: Above | 0 | 3 | 2 | 0 | 0 | 1
  Hematocrit: Unknown | 0 | 1 | 1 | 1 | 0 | 1
  Hematocrit: Below | 0 | 0 | 0 | 0 | 0 | 1
  Hematocrit: Whitin | 10 | 49 | 9 | 49 | 10 | 48
  Hematocrit: Above | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine: Unknown | 0 | 1 | 1 | 1 | 0 | 1
  Creatinine: Below | 1 | 0 | 0 | 1 | 0 | 0
  Creatinine: Whitin | 9 | 46 | 9 | 48 | 10 | 49
  Creatinine: Above | 0 | 3 | 0 | 0 | 0 | 0
  AST: Unknown | 0 | 1 | 1 | 1 | 0 | 1
  AST: Below | 0 | 0 | 0 | 0 | 0 | 0
  AST: Whitin | 10 | 49 | 8 | 48 | 9 | 48
  AST: Above | 0 | 0 | 1 | 1 | 1 | 1
  ALT: Unknown | 0 | 1 | 1 | 1 | 0 | 1
  ALT: Below | 0 | 2 | 0 | 0 | 0 | 0
  ALT: Whitin | 10 | 47 | 8 | 47 | 9 | 47
  ALT: Above | 0 | 0 | 1 | 2 | 1 | 2
  Neutrophils: Unknown | 0 | 1 | 1 | 1 | 0 | 1
  Neutrophils: Below | 1 | 5 | 1 | 7 | 0 | 2
  Neutrophils: Whitin | 9 | 41 | 8 | 42 | 10 | 46
  Neutrophils: Above | 0 | 3 | 0 | 0 | 0 | 1
  Basophils: Unknown | 0 | 1 | 1 | 1 | 0 | 1
  Basophils: Below | 0 | 0 | 0 | 0 | 0 | 0
  Basophils: Whitin | 10 | 49 | 9 | 49 | 10 | 49
  Basophils: Above | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils: Unknown | 0 | 1 | 1 | 1 | 0 | 1
  Eosinophils: Below | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils: Whitin | 8 | 46 | 8 | 46 | 10 | 47
  Eosinophils: Above | 2 | 3 | 1 | 3 | 0 | 2
  WBC: Unknown | 0 | 1 | 1 | 1 | 0 | 1
  WBC: Below | 2 | 2 | 0 | 3 | 0 | 6
  WBC: Whitin | 8 | 45 | 9 | 46 | 10 | 43
  WBC: Above | 0 | 2 | 0 | 0 | 0 | 0

12. Primary Outcome: Number of Subjects With a Response in Terms of Cluster of Differentiation 4 (CD4+) T-cells Expressing at Least Two Cytokines Including IL-2 Equal or Above the Cut-off to at Least 1, 2, 3 Antigens and to All 4 Antigens
Description: Antigen-specific CD4+ T-cells can express cluster of differentiation 40-ligand (CD40-L) and produce the cytokines Interleukin 2 (IL-2) and/or Tumor Necrosis Factor alpha (TNF-α) and/or Interferon-gamma (IFN-γ). The frequency of antigen specific CD4+T-cells was calculated as the difference between the frequency of CD4+T-cells producing at least 2 cytokines (among IFN-g, IL-2, TNF-a and/or CD40L), upon in vitro stimulation with the peptide pools derived from the antigen minus the frequency of CD4+T-cells producing at least 2 cytokines upon in vitro stimulation in medium only.A responder was a subject with an antigen-stimulated CD4+T cells response greater than or equal to the cut-off value. The same cut-off value was used for all subjects and all antigen responses post-vaccination. It was calculated from the pre-vaccination CD4+T cell responses (the frequency of antigen-stimulated CD4+T cells expressing at least two markers; i.e. all doubles) for all subjects.
Time Frame: At Day 44
Population: Analysis was performed on the According-to-Protocol cohort for Immunogenicity that included all evaluable subjects (i.e. those meeting all eligibility criteria, complying with procedures and intervals defined in protocol, with no elimination criteria during study) for whom data concerning immunogenicity outcome measures were available.
Measure: Count of Participants; unit: Participants
Arm/Group | SB732461 Non-adjuvanted_LD Group | SB732461 Non-adjuvanted_MD Group | SB732461 Non-adjuvanted_HD Group | SB732461 adjuvanted_LD Group | SB732461 adjuvanted_MD Group | SB732461 adjuvanted_HD Group
Number analyzed (Participants) | 8 | 9 | 9 | 46 | 40 | 35
Participants
  At least 1 antigen | 1 | 2 | 2 | 46 | 40 | 35
  At least 2 antigens | 0 | 1 | 2 | 46 | 38 | 34
  At least 3 antigens | 0 | 1 | 0 | 46 | 34 | 31
  All 4 antigens | 0 | 0 | 0 | 37 | 22 | 23

13. Secondary Outcome: Frequency of p17, p24, Nef and RT-specific CD4+ T-cells Expressing IL-2 and at Least Another Marker
Description: Antigen-specific CD4+ T-cells can express CD40 ligand (CD40-L) and produce the cytokines Interleukin 2 (IL-2) and/or Tumor Necrosis Factor alpha (TNF-α) and/or Interferon-gamma (IFN-γ). Frequency of CD4+ T-cells expressing markers in response to the F4co fusion protein (all antigens) was estimated by adding individual frequencies of CD4+ T-cells to each of the 4 antigens (p17, p24, Nef, RT). Results are presented as determined by Intracellular Cytokine Staining (ICS).
Time Frame: At Month 0, Day 44, Month 2, Month 6 and Month 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: CD4+ T-cells/million T-cells
Arm/Group | SB732461 Non-adjuvanted_LD Group | SB732461 Non-adjuvanted_MD Group | SB732461 Non-adjuvanted_HD Group | SB732461 adjuvanted_LD Group | SB732461 adjuvanted_MD Group | SB732461 adjuvanted_HD Group
Number analyzed (Participants) | 9 | 9 | 9 | 46 | 40 | 35
CD4+ T-cells/million T-cells
  p17, Day 0: number analyzed (Participants) | 9 | 9 | 9 | 43 | 40 | 35
  p17, Day 0 | 32.56 (46.31) | 16.78 (16.08) | 7.89 (10.86) | 17.95 (25.64) | 21.90 (44.84) | 30.60 (49.28)
  p17, Day 44: number analyzed (Participants) | 8 | 9 | 9 | 46 | 40 | 35
  p17, Day 44 | 58.25 (67.23) | 102.00 (171.17) | 57.22 (76.97) | 1724.07 (1335.80) | 696.78 (592.73) | 740.91 (637.48)
  p17, Month 2: number analyzed (Participants) | 9 | 9 | 9 | 44 | 40 | 33
  p17, Month 2 | 17.33 (28.18) | 60.11 (79.90) | 30.22 (40.38) | 1238.82 (968.59) | 517.38 (440.05) | 625.88 (525.66)
  p17, Month 6: number analyzed (Participants) | 9 | 8 | 8 | 46 | 40 | 34
  p17, Month 6 | 22.22 (28.83) | 80.50 (119.81) | 61.63 (74.83) | 762.59 (608.13) | 376.80 (291.36) | 360.32 (324.15)
  p17, Month 12: number analyzed (Participants) | 8 | 8 | 9 | 44 | 40 | 35
  p17, Month 12 | 28.50 (42.64) | 70.13 (140.50) | 25.00 (28.14) | 766.55 (620.56) | 345.55 (320.76) | 462.29 (439.06)
  p24, Day 0: number analyzed (Participants) | 9 | 9 | 9 | 43 | 40 | 35
  p24, Day 0 | 51.67 (55.49) | 27.56 (48.52) | 29.11 (43.11) | 30.60 (41.68) | 54.95 (68.53) | 52.14 (80.65)
  p24, Day 44: number analyzed (Participants) | 8 | 9 | 9 | 46 | 40 | 35
  p24, Day 44 | 47.25 (38.39) | 205.22 (375.13) | 119.22 (160.14) | 3078.59 (1694.26) | 1441.93 (1286.57) | 1446.17 (990.24)
  p24, Month 2: number analyzed (Participants) | 9 | 9 | 9 | 44 | 40 | 33
  p24, Month 2 | 31.56 (58.84) | 142.67 (138.05) | 87.22 (83.82) | 2228.00 (1255.40) | 1171.50 (1220.16) | 1120.58 (654.53)
  p24, Month 6: number analyzed (Participants) | 9 | 8 | 8 | 46 | 40 | 34
  p24, Month 6 | 53.78 (85.56) | 83.75 (122.43) | 143.63 (130.22) | 1320.63 (1002.27) | 775.63 (588.91) | 562.26 (402.53)
  p24, Month 12: number analyzed (Participants) | 8 | 8 | 9 | 44 | 40 | 35
  p24, Month 12 | 34.25 (38.37) | 74.00 (77.45) | 101.78 (108.18) | 1282.00 (819.01) | 766.55 (549.94) | 718.17 (533.47)
  Nef, Day 0: number analyzed (Participants) | 9 | 9 | 9 | 43 | 40 | 35
  Nef, Day 0 | 25.78 (45.94) | 22.00 (40.81) | 78.11 (98.18) | 40.02 (49.98) | 39.53 (59.12) | 58.97 (101.11)
  Nef, Day 44: number analyzed (Participants) | 8 | 9 | 9 | 46 | 40 | 35
  Nef, Day 44 | 52.63 (65.28) | 89.00 (81.17) | 108.22 (97.17) | 1822.50 (1553.80) | 872.83 (706.00) | 862.20 (721.64)
  Nef, Month 2: number analyzed (Participants) | 9 | 9 | 9 | 44 | 40 | 33
  Nef, Month 2 | 30.56 (55.59) | 75.67 (104.05) | 73.00 (93.10) | 1307.89 (1080.10) | 678.78 (503.13) | 713.33 (490.14)
  Nef, Month 6: number analyzed (Participants) | 9 | 8 | 8 | 46 | 40 | 34
  Nef, Month 6 | 46.67 (70.30) | 36.25 (56.89) | 38.75 (40.15) | 855.13 (901.48) | 532.80 (508.78) | 374.32 (302.71)
  Nef, Month 12: number analyzed (Participants) | 8 | 8 | 9 | 44 | 40 | 35
  Nef, Month 12 | 23.00 (36.26) | 20.75 (47.65) | 42.56 (66.95) | 722.80 (780.58) | 404.98 (364.64) | 426.34 (447.54)
  RT, Day 0: number analyzed (Participants) | 9 | 9 | 9 | 43 | 40 | 35
  RT, Day 0 | 77.44 (83.84) | 31.67 (44.13) | 21.33 (27.16) | 52.53 (109.33) | 52.85 (96.57) | 63.80 (74.44)
  RT, Day 44: number analyzed (Participants) | 8 | 9 | 9 | 46 | 40 | 35
  RT, Day 44 | 107.75 (115.20) | 250.00 (351.18) | 262.00 (327.68) | 6760.11 (3832.30) | 2787.43 (1785.69) | 2518.71 (1389.15)
  RT, Month 2: number analyzed (Participants) | 9 | 9 | 9 | 44 | 40 | 33
  RT, Month 2 | 109.22 (67.04) | 242.22 (349.31) | 209.89 (363.37) | 4731.64 (2761.73) | 2304.75 (1798.00) | 2107.61 (1107.18)
  RT, Month 6: number analyzed (Participants) | 9 | 8 | 8 | 46 | 40 | 34
  RT, Month 6 | 46.67 (61.07) | 140.75 (210.46) | 103.88 (165.37) | 3157.02 (2345.20) | 1539.85 (1100.27) | 1198.74 (748.47)
  RT, Month 12: number analyzed (Participants) | 8 | 8 | 9 | 44 | 40 | 35
  RT, Month 12 | 54.50 (59.96) | 99.38 (106.52) | 132.33 (216.98) | 2965.34 (2148.86) | 1433.63 (1020.80) | 1347.26 (988.06)

14. Secondary Outcome: Frequency of p17, p24, Nef and RT-specific CD4+ T-cells Expressing at Least 2 Immune Markers
Description: as for outcome 13
Time Frame: At Month 0, Day 44, Month 2, Month 6 and Month 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: CD4+ T-cells/million T-cells
Arm/Group | SB732461 Non-adjuvanted_LD Group | SB732461 Non-adjuvanted_MD Group | SB732461 Non-adjuvanted_HD Group | SB732461 adjuvanted_LD Group | SB732461 adjuvanted_MD Group | SB732461 adjuvanted_HD Group
Number analyzed (Participants) | 9 | 9 | 9 | 46 | 40 | 35
CD4+ T-cells/million T-cells
  p17, Day 0: number analyzed (Participants) | 9 | 9 | 9 | 43 | 40 | 35
  p17, Day 0 | 21.89 (30.92) | 5.56 (10.45) | 30.44 (63.90) | 23.58 (34.72) | 32.75 (62.91) | 39.80 (65.83)
  p17, Day 44: number analyzed (Participants) | 8 | 9 | 9 | 46 | 40 | 35
  p17, Day 44 | 59.75 (76.90) | 104.22 (146.67) | 69.67 (84.30) | 1937.11 (1457.55) | 777.68 (662.55) | 850.86 (724.32)
  p17, Month 2: number analyzed (Participants) | 9 | 9 | 9 | 44 | 40 | 33
  p17, Month 2 | 15.11 (24.79) | 65.56 (84.74) | 23.00 (30.72) | 1308.50 (1000.94) | 562.63 (473.95) | 682.70 (553.88)
  p17, Month 6: number analyzed (Participants) | 9 | 8 | 8 | 46 | 40 | 35
  p17, Month 6 | 57.78 (72.39) | 101.38 (132.38) | 94.13 (112.30) | 791.54 (636.43) | 411.95 (290.81) | 398.62 (348.32)
  p17, Month 12: number analyzed (Participants) | 8 | 8 | 9 | 44 | 40 | 35
  p17, Month 12 | 32.13 (45.05) | 101.25 (197.89) | 31.00 (36.44) | 784.57 (613.62) | 374.65 (319.92) | 501.60 (451.23)
  p24, Day 0: number analyzed (Participants) | 9 | 9 | 9 | 43 | 40 | 35
  p24, Day 0 | 46.67 (51.44) | 46.56 (78.36) | 93.56 (155.14) | 60.05 (67.01) | 77.98 (87.63) | 68.31 (100.00)
  p24, Day 44: number analyzed (Participants) | 8 | 9 | 9 | 46 | 40 | 35
  p24, Day 44 | 80.13 (47.22) | 243.00 (441.48) | 161.56 (161.44) | 3536.04 (1850.10) | 1662.85 (1462.02) | 1661.03 (1108.49)
  p24, Month 2: number analyzed (Participants) | 9 | 9 | 9 | 44 | 40 | 33
  p24, Month 2 | 49.11 (83.84) | 145.56 (179.74) | 121.89 (152.43) | 2429.89 (1309.28) | 1306.25 (1320.29) | 1253.06 (685.13)
  p24, Month 6: number analyzed (Participants) | 9 | 8 | 8 | 46 | 40 | 34
  p24, Month 6 | 53.78 (53.78) | 83.75 (122.43) | 143.63 (130.22) | 1320.63 (1002.27) | 775.63 (588.91) | 562.26 (402.53)
  p24, Month 12: number analyzed (Participants) | 8 | 8 | 9 | 44 | 40 | 35
  p24, Month 12 | 34.25 (38.37) | 74.00 (77.45) | 101.78 (108.18) | 1282.00 (819.01) | 766.55 (549.94) | 718.17 (533.47)
  Nef, Day 0: number analyzed (Participants) | 9 | 9 | 9 | 43 | 40 | 35
  Nef, Day 0 | 18.67 (36.54) | 30.00 (57.59) | 157.56 (206.05) | 52.74 (64.54) | 60.70 (91.26) | 80.51 (126.89)
  Nef, Day 44: number analyzed (Participants) | 8 | 9 | 9 | 46 | 40 | 35
  Nef, Day 44 | 61.00 (77.57) | 87.11 (64.23) | 138.44 (123.44) | 2133.76 (1825.49) | 1039.80 (830.73) | 1034.77 (836.85)
  Nef, Month 2: number analyzed (Participants) | 9 | 9 | 9 | 44 | 40 | 33
  Nef, Month 2 | 51.78 (82.87) | 69.89 (143.34) | 99.78 (123.76) | 1470.00 (1160.99) | 751.35 (521.38) | 826.45 (539.88)
  Nef, Month 6: number analyzed (Participants) | 9 | 8 | 8 | 46 | 40 | 34
  Nef, Month 6 | 66.67 (64.44) | 29.75 (46.20) | 73.75 (55.65) | 906.78 (935.03) | 574.18 (536.34) | 435.71 (293.58)
  Nef, Month 12: number analyzed (Participants) | 8 | 8 | 9 | 44 | 40 | 35
  Nef, Month 12 | 60.50 (61.35) | 45.63 (50.45) | 50.44 (54.97) | 786.23 (803.67) | 432.85 (379.08) | 485.23 (478.78)
  RT, Day 0: number analyzed (Participants) | 9 | 9 | 9 | 43 | 40 | 35
  RT, Day 0 | 158.56 (363.46) | 60.78 (71.21) | 47.22 (44.13) | 107.84 (225.52) | 81.00 (143.07) | 148.37 (346.73)
  RT, Day 44: number analyzed (Participants) | 8 | 9 | 9 | 46 | 40 | 35
  RT, Day 44 | 328.25 (556.42) | 311.00 (352.09) | 297.78 (368.77) | 7843.87 (4284.29) | 3231.88 (2077.15) | 3041.74 (1961.13)
  RT, Month 2: number analyzed (Participants) | 9 | 9 | 9 | 44 | 40 | 33
  RT, Month 2 | 365.00 (729.94) | 261.78 (385.82) | 283.56 (380.40) | 5291.91 (2921.62) | 2575.98 (1972.59) | 2471.94 (1509.43)
  RT, Month 6: number analyzed (Participants) | 9 | 8 | 8 | 46 | 40 | 34
  RT, Month 6 | 46.67 (61.07) | 140.75 (210.46) | 103.88 (165.37) | 3157.02 (2345.20) | 1539.85 (1100.27) | 1198.74 (748.47)
  RT, Month 12: number analyzed (Participants) | 8 | 8 | 9 | 44 | 40 | 35
  RT, Month 12 | 54.50 (59.96) | 99.38 (106.52) | 132.33 (216.98) | 2965.34 (2148.86) | 1433.63 (1020.80) | 1347.26 (988.06)

15. Secondary Outcome: Antibody Titers Against p17, p24, Nef, RT and F4co Antigens
Description: Anti-p17, -p24, -Nef, -RT and -F4co antibody titers were measured by Enzyme Linked Immunosorbent Assay (ELISA) and presented as geometric mean titers (GMTs).
Time Frame: At Month 0, Day 44, Month 2, Month 6 and Month 12
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | SB732461 Non-adjuvanted_LD Group | SB732461 Non-adjuvanted_MD Group | SB732461 Non-adjuvanted_HD Group | SB732461 adjuvanted_LD Group | SB732461 adjuvanted_MD Group | SB732461 adjuvanted_HD Group
Number analyzed (Participants) | 9 | 9 | 9 | 49 | 41 | 35
Titers
  Anti-p17, Day 0 | 93.5 [93.5 to 93.5] | 109.5 [76.1 to 157.4] | 93.5 [93.5 to 93.5] | 93.5 [93.5 to 93.5] | 93.5 [93.5 to 93.5] | 96.3 [90.7 to 102.1]
  Anti-p17, Day 44 | 93.5 [93.5 to 93.5] | 133.3 [76.4 to 232.7] | 104.2 [81.2 to 133.8] | 824.9 [518.6 to 1312.1] | 1416.4 [888.0 to 2259.4] | 1499.7 [872.1 to 2579.0]
  Anti-p17, Month 2: number analyzed (Participants) | 9 | 9 | 9 | 49 | 40 | 35
  Anti-p17, Month 2 | 93.5 [93.5 to 93.5] | 107.6 [77.8 to 148.9] | 93.5 [93.5 to 93.5] | 553.2 [354.8 to 862.6] | 808.2 [529.1 to 1234.5] | 1189.3 [730.5 to 1936.3]
  Anti-p17, Month 6: number analyzed (Participants) | 9 | 8 | 8 | 46 | 40 | 34
  Anti-p17, Month 6 | 93.5 [93.5 to 93.5] | 93.5 [93.5 to 93.5] | 93.5 [93.5 to 93.5] | 169.0 [128.3 to 222.7] | 167.4 [121.1 to 231.4] | 146.6 [112.7 to 190.8]
  Anti-p17, Month 12: number analyzed (Participants) | 9 | 8 | 9 | 46 | 40 | 33
  Anti-p17, Month 12 | 93.5 [93.5 to 93.5] | 93.5 [93.5 to 93.5] | 93.5 [93.5 to 93.5] | 128.0 [101.6 to 161.2] | 140.5 [109.4 to 180.5] | 133.7 [102.8 to 173.9]
  Anti-p24, Day 0 | 59.5 [59.5 to 59.5] | 64.7 [53.3 to 78.6] | 59.5 [59.5 to 59.5] | 59.5 [59.5 to 59.5] | 59.5 [59.5 to 59.5] | 62.1 [56.9 to 67.8]
  Anti-p24, Day 44 | 65.3 [52.7 to 80.8] | 120.3 [57.0 to 253.9] | 88.8 [43.1 to 183.0] | 18765.3 [14750.4 to 23872.9] | 18788.8 [15248.4 to 23151.4] | 21089.3 [16184.8 to 27480.0]
  Anti-p24, Month 2: number analyzed (Participants) | 9 | 9 | 9 | 49 | 40 | 35
  Anti-p24, Month 2 | 69.7 [48.4 to 100.2] | 97.5 [52.7 to 180.2] | 87.4 [44.6 to 171.4] | 12453.4 [9769.4 to 15874.8] | 11238.4 [8896.3 to 14197.0] | 12541.9 [9459.6 to 16628.4]
  Anti-p24, Month 6: number analyzed (Participants) | 9 | 7 | 8 | 46 | 40 | 35
  Anti-p24, Month 6 | 59.5 [59.5 to 59.5] | 59.5 [59.5 to 59.5] | 83.0 [37.8 to 182.3] | 2800.2 [2069.1 to 3789.6] | 1898.0 [1393.0 to 2586.1] | 2082.9 [1483.5 to 2924.3]
  Anti-p24, Month 12: number analyzed (Participants) | 9 | 8 | 9 | 46 | 40 | 35
  Anti-p24, Month 12 | 59.5 [59.5 to 59.5] | 59.5 [59.5 to 59.5] | 70.8 [47.4 to 105.6] | 1254.8 [917.2 to 1716.6] | 840.6 [587.7 to 1202.4] | 762.6 [561.3 to 1035.9]
  Anti-Nef, Day 0 | 116.0 [116.0 to 116.0] | 138.0 [92.4 to 206.2] | 116.0 [116.0 to 116.0] | 120.0 [112.1 to 128.4] | 129.6 [109.3 to 153.7] | 136.1 [118.4 to 156.4]
  Anti-Nef, Day 44 | 157.8 [94.2 to 264.4] | 229.2 [113.2 to 464.1] | 184.6 [85.0 to 400.9] | 27263.0 [21515.5 to 34545.9] | 20504.6 [15547.5 to 27042.3] | 26844.9 [19335.8 to 37270.1]
  Anti-Nef, Month 2: number analyzed (Participants) | 9 | 9 | 9 | 49 | 40 | 35
  Anti-Nef, Month 2 | 152.1 [81.5 to 283.8] | 185.3 [89.8 to 382.2] | 168.4 [88.5 to 320.5] | 12467.6 [9650.8 to 16106.5] | 12378.1 [9440.1 to 16230.5] | 17926.2 [13040.6 to 24642.0]
  Anti-Nef, Month 6: number analyzed (Participants) | 9 | 8 | 8 | 46 | 40 | 35
  Anti-Nef, Month 6 | 144.9 [86.8 to 241.8] | 135.4 [94.0 to 195.0] | 173.8 [66.8 to 452.5] | 2133.7 [1548.8 to 2939.4] | 1617.1 [1126.4 to 2321.4] | 2712.2 [1930.5 to 3810.2]
  Anti-Nef, Month 12: number analyzed (Participants) | 9 | 8 | 9 | 46 | 40 | 34
  Anti-Nef, Month 12 | 135.9 [94.3 to 195.9] | 154.2 [99.3 to 239.5] | 116.0 [116.0 to 116.0] | 1032.4 [716.9 to 1486.6] | 710.4 [491.2 to 1027.4] | 1330.2 [948.8 to 1865.0]
  Anti-RT, Day 0 | 62.5 [62.5 to 62.5] | 62.5 [62.5 to 62.5] | 69.1 [54.8 to 87.3] | 62.5 [62.5 to 62.5] | 64.2 [60.8 to 67.8] | 62.5 [62.5 to 62.5]
  Anti-RT, Day 44 | 62.5 [62.5 to 62.5] | 95.5 [56.5 to 161.6] | 100.1 [43.3 to 231.3] | 8979.1 [6928.2 to 11637.1] | 10019.9 [8074.8 to 12433.5] | 11812.0 [9008.8 to 15487.6]
  Anti-RT, Month 2: number analyzed (Participants) | 9 | 9 | 9 | 49 | 40 | 35
  Anti-RT, Month 2 | 76.7 [47.8 to 122.9] | 85.6 [52.8 to 138.7] | 96.5 [46.0 to 202.2] | 5761.6 [4628.7 to 7171.8] | 6543.3 [5128.8 to 8347.9] | 6959.8 [5315.5 to 9112.7]
  Anti-RT, Month 6: number analyzed (Participants) | 9 | 8 | 8 | 46 | 40 | 35
  Anti-RT, Month 6 | 71.4 [52.6 to 96.9] | 75.7 [48.2 to 118.8] | 62.5 [62.5 to 62.5] | 705.5 [567.5 to 877.0] | 902.5 [672.6 to 1211.1] | 883.9 [682.3 to 1145.0]
  Anti-RT, Month 12: number analyzed (Participants) | 9 | 8 | 9 | 46 | 40 | 35
  Anti-RT, Month 12 | 74.3 [49.9 to 110.5] | 62.5 [62.5 to 62.5] | 72.0 [51.9 to 99.9] | 462.1 [358.9 to 595.0] | 428.7 [316.1 to 581.5] | 471.1 [374.6 to 592.5]
  Anti-F4co, Month 0 | 21.0 [21.0 to 21.0] | 24.6 [17.1 to 35.4] | 21.0 [21.0 to 21.0] | 21.0 [21.0 to 21.0] | 21.0 [21.0 to 21.0] | 21.5 [20.5 to 22.4]
  Anti-F4co, Day 44 | 23.8 [17.8 to 31.8] | 42.1 [18.7 to 94.9] | 42.7 [16.4 to 111.7] | 7027.2 [5768.4 to 8560.6] | 11151.6 [9207.1 to 13506.9] | 12359.6 [9291.4 to 16441.0]
  Anti-F4co, Month 2: number analyzed (Participants) | 9 | 9 | 9 | 49 | 40 | 35
  Anti-F4co, Month 2 | 26.1 [18.6 to 36.5] | 34.7 [18.3 to 65.8] | 31.5 [15.2 to 65.1] | 4770.3 [3900.0 to 5834.9] | 4607.8 [3701.8 to 5735.4] | 5438.7 [4126.5 to 7168.2]
  Anti-F4co, Month 6: number analyzed (Participants) | 9 | 8 | 8 | 46 | 41 | 35
  Anti-F4co, Month 6 | 22.9 [18.7 to 28.0] | 25.5 [18.9 to 34.6] | 31.0 [12.3 to 77.8] | 1303.1 [1065.2 to 1594.2] | 1081.4 [813.9 to 1436.8] | 1081.4 [780.0 to 1499.3]
  Anti-F4co, Month 12: number analyzed (Participants) | 9 | 8 | 9 | 46 | 41 | 35
  Anti-F4co, Month 12 | 25.1 [16.6 to 38.1] | 23.6 [17.9 to 31.2] | 33.1 [17.9 to 61.5] | 790.7 [633.4 to 987.0] | 1154.0 [839.3 to 1586.7] | 837.5 [605.2 to 1158.9]

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period; Unsolicited AEs: during the 30-day (Days 0-29) post-vaccination period; SAEs: during the entire study period (from Month 0 up to Month 12).
Arm/Group | SB732461 Non-adjuvanted_LD Group | SB732461 Non-adjuvanted_MD Group | SB732461 Non-adjuvanted_HD Group | SB732461 adjuvanted_LD Group | SB732461 adjuvanted_MD Group | SB732461 adjuvanted_HD Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/50 | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 2/50 | 2/50 | 2/50
Other Adverse Events (participants affected / at risk) | 8/10 | 7/10 | 9/10 | 50/50 | 50/50 | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB732461 Non-adjuvanted_LD Group (N=10) | SB732461 Non-adjuvanted_MD Group (N=10) | SB732461 Non-adjuvanted_HD Group (N=10) | SB732461 adjuvanted_LD Group (N=50) | SB732461 adjuvanted_MD Group (N=50) | SB732461 adjuvanted_HD Group (N=50)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Henoch-schonlein purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB732461 Non-adjuvanted_LD Group (N=10) | SB732461 Non-adjuvanted_MD Group (N=10) | SB732461 Non-adjuvanted_HD Group (N=10) | SB732461 adjuvanted_LD Group (N=50) | SB732461 adjuvanted_MD Group (N=50) | SB732461 adjuvanted_HD Group (N=50)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 9 (11) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 3 (3)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 14 (19) | 23 (35) | 25 (34)
Fatigue (General disorders) | 5 (6) | 5 (7) | 6 (9) | 41 (67) | 47 (71) | 46 (77)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (3) | 23 (29) | 21 (24) | 17 (21)
Hangover (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 4 (8) | 5 (5) | 43 (78) | 42 (65) | 41 (65)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 3 (3) | 28 (35) | 28 (33) | 26 (34)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 3 (3) | 2 (2)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 5 (6) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 2 (2) | 31 (45) | 35 (52) | 36 (52)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 3 (4) | 1 (2) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 4 (4) | 3 (4)
Pain (General disorders) | 3 (5) | 2 (2) | 5 (6) | 49 (96) | 50 (98) | 50 (97)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (4)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 30 (34) | 29 (32) | 26 (29)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Stress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 13 (20) | 18 (25) | 19 (22)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2007-10-08): https://cdn.clinicaltrials.gov/large-docs/12/NCT00434512/Prot_000.pdf
  • Statistical Analysis Plan (2008-09-26): https://cdn.clinicaltrials.gov/large-docs/12/NCT00434512/SAP_001.pdf